CLINICAL TRIAL: NCT07255768
Title: Comparison of the Efficacy of Pericapsular Nerve Group Block Alone Versus Pericapsular Nerve Group Block Combined With Superior Cluneal and Superior Gluteal Nerve Blocks in Patients Undergoing Hip Surgery: A Prospective Randomized Clinical Study
Brief Title: Comparison of the Efficacy of Pericapsular Nerve Group Block Alone Versus Pericapsular Nerve Group Block Combined With Superior Cluneal and Superior Gluteal Nerve Blocks in Patients Undergoing Hip Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PENGHip
Record Dates: First submitted 2025-11-16; First posted 2025-12-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis; Osteonecrosis of the Femoral Head; Avascular Necrosis of Femur Head; Dysplasia of Hip Joint; Hip Surgeries
MeSH Terms: conditions — Osteoarthritis, Hip; Legg-Calve-Perthes Disease; Femur Head Necrosis | interventions — Bupivacaine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of PENG Block (Active Comparator): Patients will be brought to the operating room one hour before surgery, and no premedication will be administered prior to their arrival. Before performing the PENG block, patients will be placed in the supine position. The ultrasound probe will be positioned in the transverse plane medial and caudal to the anterior superior iliac spine, and the anterior inferior iliac spine, iliopubic eminence, and psoas tendon will be identified. Using an in-plane technique, the needle will be advanced from lateral to medial and positioned between the psoas tendon and the periosteum. After negative aspiration, 15 mL of 0.25% bupivacaine will be administered.
  Interventions: Drug: 15 ml Bupivacaine Hcl 0.25% injection; Drug: 20 mL bupivacaine 0.25% injection
- Application of PENG Block together with Superior Cluneal and Superior Gluteal Nerve Blocks (Active Comparator): All patients will receive a PENG block, and in addition:
  The superior cluneal nerve block will be performed at the level of the posterior iliac crest under ultrasound guidance, along the course of the nerve, using 10 mL of 0.25% bupivacaine.
  The superior gluteal nerve block will be administered in the lateral decubitus position under ultrasound guidance, with 10 mL of 0.25% bupivacaine injected between the gluteal muscles along the trajectory of the nerve.
  Interventions: Drug: 20 mL bupivacaine 0.25% injection

INTERVENTIONS:
Drug: 15 ml Bupivacaine Hcl 0.25% injection — For PENG Block, 15 mL of 0.25% bupivacaine will be administered.
  Arms: Application of PENG Block
Drug: 20 mL bupivacaine 0.25% injection — After performing PENG; 10 mL of 0.25% bupivacaine will be administered for each superior cluneal nerve block and superior gluteal nerve block

SUMMARY:
In the clinic, total hip arthroplasty is a frequently performed surgical procedure that often results in moderate to severe postoperative pain. Multimodal analgesia approaches are commonly preferred for managing this pain, and in recent years, nerve blocks targeting pelvic innervation have become increasingly prominent. Among these, the Pericapsular Nerve Group (PENG) block has gained attention for providing effective analgesia by targeting the nerves responsible for the anterior innervation of the hip capsule. However, when used alone, the PENG block may be insufficient for controlling posterior hip pain and may not provide complete analgesia.

In this context, adding blocks targeting the superior cluneal nerve and the superior gluteal nerve-both of which contribute to the sensory innervation of the posterior hip region-has been proposed to enhance the analgesic effect when combined with the PENG block. Superior cluneal and superior gluteal nerve blocks have recently been described in anatomical and clinical studies, and by affecting the structures contributing sensory input to the posterior hip capsule, they hold significant potential for improving pain management.

In this study, the investigators aimed to evaluate the contribution of superior cluneal and superior gluteal nerve blocks, when added to the PENG block, to perioperative analgesia in patients undergoing total hip arthroplasty. The investigators sought to comparatively investigate whether this combination offers superior outcomes compared with the PENG block alone. It was hypothesized that combined nerve blocks may provide similar or improved recovery scores, lower pain scores, reduced opioid consumption, and enhanced analgesic efficacy without affecting the degree of motor blockade.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Age between 18 and 80 years
* ASA physical status I, II, or III
* Male or female patients

Exclusion Criteria:

* Refusal to participate in the study
* Allergy to the medications to be used
* History of severe cardiac, renal, or hepatic disease
* Presence of neurological deficits or neuropathy
* History of anticoagulant use
* Previous surgery in the inguinal or suprainguinal region
* Pregnancy
* Chronic opioid use at home
* History of spinal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
QoR-15 (Quality of Recovery-15) questionnaire | 24th and 48th postoperative hour
  The primary outcome measure will be the QoR-15 (Quality of Recovery-15) questionnaire administered at the 24th postoperative hour. QoR-15 is a validated 15-item short survey assessing patients' postoperative physical comfort, emotional state, level of independence, pain control, and overall well-being. The total score obtained will be used to compare the overall quality of recovery between groups. The same questionnaire will be repeated at the 48th postoperative hour.

SECONDARY OUTCOMES:
Quadriceps Motor Block Assessment | It will be assessed at the 4th, 8th, 12th, and 24th postoperative hours.
  Motor block will be assessed using the following 3-point scale:
  0 = Normal strength (dorsiflexion against gravity and resistance)
  1. = Paresis (dorsiflexion against gravity only, not against resistance)
  2. = Paralysis (dorsiflexion not possible)
Motor Block Assessment at the Tibialis Anterior Muscle for the Sciatic Nerve | It will be assessed at the 4th, 8th, 12th, and 24th postoperative hours.
  Motor block will be assessed using the following 3-point scale:
  0 = Normal strength (dorsiflexion against gravity and resistance)
  1. = Paresis (dorsiflexion against gravity only, not against resistance)
  2. = Paralysis (dorsiflexion not possible)
Fentanyl consumption | The first 24 postoperative hours
  Fentanyl consumption will be recorded via the PCA device during the postoperative intervals of 0-4, 4-8, and 8-24 hours. Total opioid consumption will be calculated at the 24th postoperative hour.
VAS pain scores | The first 24 postoperative hours
  VAS pain scores will be assessed at the 1st, 2nd, 4th, 8th, 12th, and 24th postoperative hours, both at rest and during movement. The region where the patient experiences the most intense pain will be recorded as either the anterior or posterior hip.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)